CLINICAL TRIAL: NCT02799303
Title: A Randomized Clinical Trial Comparing the Efficacy of MRI Versus PSA for Prostate Cancer Screening: The MVP Study (MRI vs PSA)
Brief Title: MRI Versus PSA in Prostate Cancer Screening
Acronym: MVP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Robert Nam, Professor of Surgery, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 130-2016
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
Keywords: screening; biopsy; magnetic resonance imaging; prostate specific antigen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Intervention not a drug/biologic.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi-parametric MRI (Experimental): Patients from the general population without history of previous prostate biopsy will be allocated to receive mpMRI in order to evaluate for risk of prostate cancer.
  Interventions: Device: Multi-parametric MRI
- PSA Only (Active Comparator): Patients from the general population without history of previous prostate biopsy will be allocated to receive serum PSA testing in order to evaluate for risk of prostate cancer.
  Patients with a serum PSA level less than 4.0 ng/mL will be managed expectantly with results provided to their primary care physician.
  Interventions: Other: PSA testing

INTERVENTIONS:
Device: Multi-parametric MRI — Non contrast magnetic resonance imaging using T1/T2 weighting, DWI and ADC will be performed. MRI images will be reviewed by a single uro-radiologist and assessed using the PiRADs standards.
  Arms: Multi-parametric MRI
Other: PSA testing — Serum prostate specific antigen (PSA) testing will be performed using a standardized laboratory assay.
  Arms: PSA Only

SUMMARY:
In this open randomized controlled trial, we seek to study whether prostate cancer screening using multiparametric prostate magnetic resonance imaging (mpMRI) improves the detection rate of clinically-significant prostate cancer (defined as Gleason score ≥7 on prostate biopsy) compared with prostate cancer screening using prostate-specific antigen (PSA).

The current paradigm of prostate cancer screening relies upon an initial PSA blood test, with subsequent investigations driven by the serum PSA level. This model has proven highly controversial due to the inability of PSA level to discern between indolent and aggressive forms of prostate cancer. As a result, numerous government-sponsored bodies have recommended against PSA screening. Evidence suggests that prostate cancer screening has led to an increased proportion of men being diagnosed with potentially curable prostate cancer. However, due to the inability of the PSA level to accurately distinguish patients with indolent and lethal forms of prostate cancer, it has led to a significant rate of over-diagnosis of indolent disease. Magnetic resonance imaging has been gaining an increasingly large role in the management of patients with clinically-localized prostate cancer including diagnosis in patients with abnormal PSA levels, monitoring of patients on active surveillance and staging prior to definitive interventions. MRI-based prostate cancer risk assessment has been shown to better distinguish between clinically-significant and insignificant tumors than PSA test. Therefore, a randomized controlled trial of MRI-based prostate cancer screening and PSA-based prostate cancer screening is warranted.

DETAILED DESCRIPTION:
BACKGROUND AND RATONALE:

Prostate cancer is the most common non-cutaneous malignancy and the third leading cause of cancer death among men in Canada1. In 1987, prostate specific antigen was introduced for prostate cancer screening2. Widespread adoption of PSA screening resulted in a significantly increased number of incident cases and a significantly reduced number of cases of metastatic disease at presentation3. Coinciding with the introduction of PSA testing, prostate cancer mortality has decreased approximately 40% from an epidemiologic perspective4. Approximately 45-70% of the decline in mortality is attributable to PSA-based prostate cancer screening5. Several studies have examined whether screening for prostate cancer using the PSA test improves overall and prostate cancer mortality. In particular, two large randomized studies in the U.S. and Europe have been conducted to evaluate this. Recently, the U.S. Preventative Services Task Force (USPSTF) reviewed these and all studies to evaluate whether PSA should be used as a screening test.

Current Recommendations for PSA Screening from the USPSTF

The USPSTF makes recommendations regarding the effectiveness of screening tests for asymptomatic patients after assessing the evidence regarding benefits and harms of an intervention. The most recent USPSTF guidelines regarding prostate cancer were published in 20126.

The first component of the USPSTF assessment is an evaluation of the benefits of early detection and treatment of prostate cancer. The review panel drew on two large randomized controlled trials which have been conducted to assess the effect of PSA-based prostate cancer screening on prostate cancer mortality: the European Randomized Study of Screening for Prostate Cancer (ERSPC)7 and the U.S.-based Prostate, Lung, Colorectal and Ovarian (PLCO) Cancer Screening Trial8. In their recommendation the guideline panel do not consider significant differences between the trials, in large part due to the fact that PSA had been widely adopted in the US during the study interval while it did not have such uptake in Europe. As a result, there are concerns that the trial did not compare screening to no screening and that the trial would be unlikely to find a benefit even if a significant one existed9. Regardless, the panel concluded that prostate cancer screening resulted in the avoidance of 0 to 1 prostate cancer deaths per 1000 men screened6, a minimal benefit.

The second component of the guideline panel's assessment focused on potential harms of early detection and treatment. They found evidence of significant harm due to false-positive PSA results which confer a risk of psychological harm in addition to medical evaluation including biopsy6. Further, they considered there to be, at minimum, a small harm associated with prostate biopsy due to pain, bleeding and infectious risk. The panel also concluded that there was significant evidence of at least moderate overdiagnosis and resultant overtreatment among patients undergoing PSA-based screening.

Due to a perceived lack of benefit and presence of significant harms, the USPSTF concluded, with moderate certainty, that the benefit of PSA-based screening did not outweigh the harms and thus recommended against PSA-based screening for prostate cancer6.

A major limitation of this task force was that they received no input from experts in prostate cancer in order to minimize bias. While this may improve the objectivity of the review, many aspects of understanding prostate cancer were lost. In response to these recommendations, the American Society of Clinical Oncology (ASCO) - the largest oncology association in North America, developed a consensus statement to address the USPSTF recommendations.

ASCO Provisional Clinical Opinion in Prostate Cancer Screening

The ASCO provisional clinical opinion on prostate cancer screening using PSA-testing was based on an Agency for Healthcare Research and Quality systematic review10. Despite drawing on the same data as the USPSTF, this panel concluded that men with a longer life expectancy (greater than 10 years) may benefit from prostate cancer screening using PSA-testing11. In men with a shorter life expectancy, PSA testing was discouraged. Unlike the USPSTF, the ASCO panel placed greater weight on the results of the ERSPC, demonstrating a significant reduction in the risk of prostate cancer death for men undergoing prostate cancer screening. They noted similar harms as the USPSTF, namely false-positive results and prostate biopsy complications.

Since the publication of this opinion, further data has become available which indicates that the relative reduction in prostate cancer death from PSA-based screening may be larger than previously estimated. The most mature data from the ERSPC has 13 years of follow up12. Based on these data, the absolute risk reduction in prostate cancer mortality from PSA screening was 0.11 per 1000 person years or 1.28 per 1000 men randomized. This risk reduction has increased with increasing duration of follow up. Additional analysis has shown an absolute risk reduction of metastatic disease was 3.1 per 1000 men randomized13. In a subgroup of the ERSPC with longer follow-up, the absolute risk reduction in prostate cancer mortality was 4.0 per 1000 men randomized14. This corresponds to a number needed to screen of 293 and number needed to diagnose of 12 in order to prevent one prostate cancer death.

Underdiagnosis of Prostate Cancer with PSA

In addition to harms of biopsy and intervention, the primary concern regarding PSA-based prostate cancer screening is the inability to distinguish between patients with indolent and aggressive forms of the disease. Prostate cancer screening programs have traditionally used a serum PSA cut-off of 4.0 ng/mL to indicate abnormality. However, many men with PSA values in excess of 4.0 ng/mL do not have prostate cancer, and even fewer have clinically significant prostate cancer. Further, up to 25% of men with PSA levels less than 4.0 ng/mL will be found to have high-grade prostate cancer, if subject to biopsy15. Thus PSA-based prostate cancer screening lacks both sensitivity and specificity to identify men with aggressive prostate cancer. As a result, in addition to significant overdiagnosis and overtreatment which has been well recognized, there is a risk for underdiagnosis.

Due to the USPSTF recommendations against PSA-based prostate cancer screening, there has been a significant decrease in PSA testing being performed by primary care physicians16. It is predicted that complete discontinuation of PSA-based screening would result in the prevention of overdiagnosis for 710,000 to 1,120,000 men in the United States over a 12 year period17. However, it would result in 36,000 to 57,000 preventable deaths due to prostate cancer over the same time period. Thus, improved methods for prostate cancer screening may allow for a diminishment in overdiagnosis while avoiding preventable deaths from prostate cancer.

Magnetic Resonance Imaging (MRI) of The Prostate

Multiparametric prostate magnetic resonance imaging (mpMRI) has an increasingly large role in the management of patients with clinically-localized prostate cancer. MpMRI was initially used as a staging test in patients with prostate cancer18. Despite the use of what would now be considered obsolete technologies, Bezzi et al. demonstrated in 1988 that MRI could identify nodal metastases with an accuracy of 88% and could distinguish disease localized to the prostate from that invading beyond the capsule with an accuracy of 78% among patients undergoing prostatectomy18. Since that time, there has been a migration in the use of MRI earlier in the disease process.

In the realm of prostate cancer treatment, MRI is used for the monitoring of patients on active surveillance following a prostate cancer diagnosis as a means of reducing prostate biopsies, with their incumbent risks19,20. When performed in the evaluation of patients with elevated PSA levels with previous negative prostate biopsy, mpMRI has been shown to identify clinically significant prostate cancers which would have been otherwise missed by routine systematic biopsy21. The use of MRI and ultrasound fusion imaging in the targeting of prostate biopsy has increased detection of clinically significant prostate cancer while limiting the diagnosis of clinically insignificant prostate cancer22.

Among men with an abnormal PSA who have never undergone a prostate biopsy, mpMRI demonstrated promise in both the detection and exclusion of prostate cancer, using an extensive prostate mapping biopsy (median 41 cores) as the referent23: the AUC was 0.27 (95% CI 0.65-0.79). In a multivariable analysis of an independent cohort including age, family history, prior 5-alpha reductase inhibitor use, digital rectal examination findings, PSA level, PSA density, and MRI score, only MRI score was predictive of clinically significant (Gleason score ≥7) prostate cancer among men without a history of previous prostate biopsy (adjusted OR 40.2, p=0.01)24.

While historically prostate MRI has required the use of an endorectal coil25, recent advances in MRI technology have obviated the need for the coil26, thus reducing the cost and burden of the imaging.

Pilot Study to Examining the Feasibility of MRI Prostate Cancer Screening

We recently conducted a pilot study assessing the feasibility of mpMRI as an initial prostate cancer screening test27. Following a newspaper based call for volunteers, we had 319 men present for possible inclusion in this study. Of these, 120 were eligible, 50 were enrolled due to limitations in funding, and 47 completed the study protocol. Serum PSA testing, mpMRI, digital rectal examination, and systematic (+/- targeted) prostate biopsies were performed on all men.

Prostate cancer was identified in 18 of 47 men (38.3%). MpMRI (AUC 0.81, 95% CI 0.67-0.94) significantly outperformed PSA (AUC 0.67, 95% CI 0.52-0.84) in the prediction of prostate cancer. In multivariable analyses including age, digital rectal examination findings, PSA and MRI score, mpMRI was the only significant predictor for the presence of prostate cancer (adjusted OR 2.7, 95% CI 1.4-5.4). These findings persisted when we sought to predict only clinically significant prostate cancer (Gleason ≥7; adjusted OR 3.5, 95% CI 1.5-8.3).

To better evaluate the use of mpMRI in prostate, a large, randomized study comparing the efficacy of mpMRI in diagnosing clinically significant, aggressive prostate cancer, compared to conventional PSA screening will be required.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 50 years old
* life expectancy greater than or equal to 10 years, according to the clinical judgement of study investigators

Exclusion Criteria:

* history of previous prostate biopsy
* PSA level measurement within 3 years of recruitment date
* abnormal digital rectal examination of the prostate consistent with prostate cancer
* history of prostate cancer in one or more first-degree relatives diagnosed at less than 50 years of age
* lower urinary tract voiding symptoms (IPSS greater than or equal to 8)
* prior or current use of 5-alpha reductase inhibitor medications (finasteride or dutasteride)
* patient unable to communicate in English in order to give proper informed consent
* claustrophobia or other medical indication which would preclude MRI
* any medical condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1010 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Clinically-significant prostate cancer | Within 3 years of randomization
  Gleason score greater than or equal to 7 on TRUS prostate biopsy

SECONDARY OUTCOMES:
Clinically-insignificant prostate cancer | Within 3 years of randomizations
  Gleason score equal to 6 on TRUS prostate biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nam, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stamey TA, Yang N, Hay AR, McNeal JE, Freiha FS, Redwine E. Prostate-specific antigen as a serum marker for adenocarcinoma of the prostate. N Engl J Med. 1987 Oct 8;317(15):909-16. doi: 10.1056/NEJM198710083171501. PMID 2442609
- [Background] Etzioni R, Gulati R, Falcon S, Penson DF. Impact of PSA screening on the incidence of advanced stage prostate cancer in the United States: a surveillance modeling approach. Med Decis Making. 2008 May-Jun;28(3):323-31. doi: 10.1177/0272989X07312719. Epub 2008 Mar 4. PMID 18319508
- [Background] Barocas DA, Mallin K, Graves AJ, Penson DF, Palis B, Winchester DP, Chang SS. Effect of the USPSTF Grade D Recommendation against Screening for Prostate Cancer on Incident Prostate Cancer Diagnoses in the United States. J Urol. 2015 Dec;194(6):1587-93. doi: 10.1016/j.juro.2015.06.075. Epub 2015 Jun 15. PMID 26087383
- [Background] Etzioni R, Tsodikov A, Mariotto A, Szabo A, Falcon S, Wegelin J, DiTommaso D, Karnofski K, Gulati R, Penson DF, Feuer E. Quantifying the role of PSA screening in the US prostate cancer mortality decline. Cancer Causes Control. 2008 Mar;19(2):175-81. doi: 10.1007/s10552-007-9083-8. Epub 2007 Nov 20. PMID 18027095
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for prostate cancer: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2012 Jul 17;157(2):120-34. doi: 10.7326/0003-4819-157-2-201207170-00459. PMID 22801674
- [Background] Schroder FH, Hugosson J, Roobol MJ, Tammela TL, Ciatto S, Nelen V, Kwiatkowski M, Lujan M, Lilja H, Zappa M, Denis LJ, Recker F, Berenguer A, Maattanen L, Bangma CH, Aus G, Villers A, Rebillard X, van der Kwast T, Blijenberg BG, Moss SM, de Koning HJ, Auvinen A; ERSPC Investigators. Screening and prostate-cancer mortality in a randomized European study. N Engl J Med. 2009 Mar 26;360(13):1320-8. doi: 10.1056/NEJMoa0810084. Epub 2009 Mar 18. PMID 19297566
- [Background] Andriole GL, Crawford ED, Grubb RL 3rd, Buys SS, Chia D, Church TR, Fouad MN, Gelmann EP, Kvale PA, Reding DJ, Weissfeld JL, Yokochi LA, O'Brien B, Clapp JD, Rathmell JM, Riley TL, Hayes RB, Kramer BS, Izmirlian G, Miller AB, Pinsky PF, Prorok PC, Gohagan JK, Berg CD; PLCO Project Team. Mortality results from a randomized prostate-cancer screening trial. N Engl J Med. 2009 Mar 26;360(13):1310-9. doi: 10.1056/NEJMoa0810696. Epub 2009 Mar 18. PMID 19297565
- [Background] Gulati R, Tsodikov A, Wever EM, Mariotto AB, Heijnsdijk EA, Katcher J, de Koning HJ, Etzioni R. The impact of PLCO control arm contamination on perceived PSA screening efficacy. Cancer Causes Control. 2012 Jun;23(6):827-35. doi: 10.1007/s10552-012-9951-8. Epub 2012 Apr 10. PMID 22488488
- [Background] Basch E, Oliver TK, Vickers A, Thompson I, Kantoff P, Parnes H, Loblaw DA, Roth B, Williams J, Nam RK. Screening for prostate cancer with prostate-specific antigen testing: American Society of Clinical Oncology Provisional Clinical Opinion. J Clin Oncol. 2012 Aug 20;30(24):3020-5. doi: 10.1200/JCO.2012.43.3441. Epub 2012 Jul 16. PMID 22802323
- [Background] Schroder FH, Hugosson J, Roobol MJ, Tammela TL, Zappa M, Nelen V, Kwiatkowski M, Lujan M, Maattanen L, Lilja H, Denis LJ, Recker F, Paez A, Bangma CH, Carlsson S, Puliti D, Villers A, Rebillard X, Hakama M, Stenman UH, Kujala P, Taari K, Aus G, Huber A, van der Kwast TH, van Schaik RH, de Koning HJ, Moss SM, Auvinen A; ERSPC Investigators. Screening and prostate cancer mortality: results of the European Randomised Study of Screening for Prostate Cancer (ERSPC) at 13 years of follow-up. Lancet. 2014 Dec 6;384(9959):2027-35. doi: 10.1016/S0140-6736(14)60525-0. Epub 2014 Aug 6. PMID 25108889
- [Background] Schroder FH, Hugosson J, Carlsson S, Tammela T, Maattanen L, Auvinen A, Kwiatkowski M, Recker F, Roobol MJ. Screening for prostate cancer decreases the risk of developing metastatic disease: findings from the European Randomized Study of Screening for Prostate Cancer (ERSPC). Eur Urol. 2012 Nov;62(5):745-52. doi: 10.1016/j.eururo.2012.05.068. Epub 2012 Jun 7. PMID 22704366
- [Background] Hugosson J, Carlsson S, Aus G, Bergdahl S, Khatami A, Lodding P, Pihl CG, Stranne J, Holmberg E, Lilja H. Mortality results from the Goteborg randomised population-based prostate-cancer screening trial. Lancet Oncol. 2010 Aug;11(8):725-32. doi: 10.1016/S1470-2045(10)70146-7. Epub 2010 Jul 2. PMID 20598634
- [Background] Thompson IM, Pauler DK, Goodman PJ, Tangen CM, Lucia MS, Parnes HL, Minasian LM, Ford LG, Lippman SM, Crawford ED, Crowley JJ, Coltman CA Jr. Prevalence of prostate cancer among men with a prostate-specific antigen level < or =4.0 ng per milliliter. N Engl J Med. 2004 May 27;350(22):2239-46. doi: 10.1056/NEJMoa031918. PMID 15163773
- [Background] Zavaski ME, Meyer CP, Sammon JD, Hanske J, Gupta S, Sun M, Trinh QD. Differences in Prostate-Specific Antigen Testing Among Urologists and Primary Care Physicians Following the 2012 USPSTF Recommendations. JAMA Intern Med. 2016 Apr;176(4):546-7. doi: 10.1001/jamainternmed.2015.7901. No abstract available. PMID 26857148
- [Background] Gulati R, Tsodikov A, Etzioni R, Hunter-Merrill RA, Gore JL, Mariotto AB, Cooperberg MR. Expected population impacts of discontinued prostate-specific antigen screening. Cancer. 2014 Nov 15;120(22):3519-26. doi: 10.1002/cncr.28932. Epub 2014 Jul 25. PMID 25065910
- [Background] Bezzi M, Kressel HY, Allen KS, Schiebler ML, Altman HG, Wein AJ, Pollack HM. Prostatic carcinoma: staging with MR imaging at 1.5 T. Radiology. 1988 Nov;169(2):339-46. doi: 10.1148/radiology.169.2.3174982.
- [Background] Recabal P, Ehdaie B. The role of MRI in active surveillance for men with localized prostate cancer. Curr Opin Urol. 2015 Nov;25(6):504-9. doi: 10.1097/MOU.0000000000000221. PMID 26372037
- [Background] Henderson DR, de Souza NM, Thomas K, Riches SF, Morgan VA, Sohaib SA, Dearnaley DP, Parker CC, van As NJ. Nine-year Follow-up for a Study of Diffusion-weighted Magnetic Resonance Imaging in a Prospective Prostate Cancer Active Surveillance Cohort. Eur Urol. 2016 Jun;69(6):1028-33. doi: 10.1016/j.eururo.2015.10.010. Epub 2015 Oct 21. PMID 26482887
- [Background] Vourganti S, Rastinehad A, Yerram N, Nix J, Volkin D, Hoang A, Turkbey B, Gupta GN, Kruecker J, Linehan WM, Choyke PL, Wood BJ, Pinto PA. Multiparametric magnetic resonance imaging and ultrasound fusion biopsy detect prostate cancer in patients with prior negative transrectal ultrasound biopsies. J Urol. 2012 Dec;188(6):2152-2157. doi: 10.1016/j.juro.2012.08.025. Epub 2012 Oct 18. PMID 23083875
- [Background] Meng X, Rosenkrantz AB, Mendhiratta N, Fenstermaker M, Huang R, Wysock JS, Bjurlin MA, Marshall S, Deng FM, Zhou M, Melamed J, Huang WC, Lepor H, Taneja SS. Relationship Between Prebiopsy Multiparametric Magnetic Resonance Imaging (MRI), Biopsy Indication, and MRI-ultrasound Fusion-targeted Prostate Biopsy Outcomes. Eur Urol. 2016 Mar;69(3):512-7. doi: 10.1016/j.eururo.2015.06.005. Epub 2015 Jun 22. PMID 26112001
- [Background] Abd-Alazeez M, Kirkham A, Ahmed HU, Arya M, Anastasiadis E, Charman SC, Freeman A, Emberton M. Performance of multiparametric MRI in men at risk of prostate cancer before the first biopsy: a paired validating cohort study using template prostate mapping biopsies as the reference standard. Prostate Cancer Prostatic Dis. 2014 Mar;17(1):40-6. doi: 10.1038/pcan.2013.43. Epub 2013 Oct 15. PMID 24126797
- [Background] Weaver JK, Kim EH, Vetter JM, Fowler KJ, Siegel CL, Andriole GL. Presence of Magnetic Resonance Imaging Suspicious Lesion Predicts Gleason 7 or Greater Prostate Cancer in Biopsy-Naive Patients. Urology. 2016 Feb;88:119-24. doi: 10.1016/j.urology.2015.10.023. Epub 2015 Nov 3. PMID 26545849
- [Background] Turkbey B, Bernardo M, Merino MJ, Wood BJ, Pinto PA, Choyke PL. MRI of localized prostate cancer: coming of age in the PSA era. Diagn Interv Radiol. 2012 Jan-Feb;18(1):34-45. doi: 10.4261/1305-3825.DIR.4478-11.1. Epub 2011 Sep 16. PMID 21922459
- [Background] Barentsz JO, Richenberg J, Clements R, Choyke P, Verma S, Villeirs G, Rouviere O, Logager V, Futterer JJ; European Society of Urogenital Radiology. ESUR prostate MR guidelines 2012. Eur Radiol. 2012 Apr;22(4):746-57. doi: 10.1007/s00330-011-2377-y. Epub 2012 Feb 10. PMID 22322308
- [Background] Nam RK, Wallis CJ, Stojcic-Bendavid J, Milot L, Sherman C, Sugar L, Haider MA. A Pilot Study to Evaluate the Role of Magnetic Resonance Imaging for Prostate Cancer Screening in the General Population. J Urol. 2016 Aug;196(2):361-6. doi: 10.1016/j.juro.2016.01.114. Epub 2016 Feb 13. PMID 26880413
- [Background] Puech P, Rouviere O, Renard-Penna R, Villers A, Devos P, Colombel M, Bitker MO, Leroy X, Mege-Lechevallier F, Comperat E, Ouzzane A, Lemaitre L. Prostate cancer diagnosis: multiparametric MR-targeted biopsy with cognitive and transrectal US-MR fusion guidance versus systematic biopsy--prospective multicenter study. Radiology. 2013 Aug;268(2):461-9. doi: 10.1148/radiol.13121501. Epub 2013 Apr 11. PMID 23579051
- [Background] Chou R, Dana T, Bougatsos C, Fu R, Blazina I, Gleitsmann K, Rugge JB. Treatments for Localized Prostate Cancer: Systematic Review to Update the 2002 U.S. Preventive Services Task Force Recommendation [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2011 Oct. Report No.: 12-05161-EF-1. Available from http://www.ncbi.nlm.nih.gov/books/NBK82315/ PMID 22171386
- [Derived] Nam R, Patel C, Milot L, Hird A, Wallis C, Macinnis P, Singh M, Emmenegger U, Sherman C, Haider MA. Prostate MRI versus PSA screening for prostate cancer detection (the MVP Study): a randomised clinical trial. BMJ Open. 2022 Nov 8;12(11):e059482. doi: 10.1136/bmjopen-2021-059482. PMID 36351725